CLINICAL TRIAL: NCT02197689
Title: Mobile Intelligent Personal Medication Management Platform
Brief Title: A Trial for a Personalized Medication Management Platform to Improve Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Taipei Veterans General Hospital, Taiwan (Other Government); China Medical University, Taiwan (Other); Taipei Medical University WanFang Hospital (Other); National Yang Ming Chiao Tung University (Other); National Chung Cheng University (Other); National Tsing Hua University, HsinChu City, Taiwan (Unknown); National Taiwan University (Other); Hwa Hsia Institute of Technology, New Taipei City, Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NSC 99-2218-E-038-001
Record Dates: First submitted 2014-07-17; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-06

CONDITIONS: Patients Take Medicine
Keywords: Personalized Medication Management; Medication Adherence; SMS Medication Reminder
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS Medication Reminder (Experimental): 763 patients were assigned to experimental group
  Interventions: Device: Personalized Medication Management Platform for SMS Reminder
- No SMS Reminder (No Intervention): 435 patients were assigned to control group as no SMS reminder

INTERVENTIONS:
Device: Personalized Medication Management Platform for SMS Reminder — The Personalized Medication Management Platform was developed by investigators that integrated with Hospital Information System (HIS) to collect the prescription information of patients and automatically send SMS to remind
  Arms: SMS Medication Reminder

SUMMARY:
Taiwan has attracted much attention for its National Health Insurance (NHI) and healthcare system around the world with many countries in Europe and the United States using it as a benchmark. However, increasing medication costs over the past two years account for more than 25% of total expenditure, surpassing every OECD member and mounting increasing pressure on the NHI. Nevertheless, patient medication adherence is relatively low. Thus, the investigators assessed the effectiveness of a personalized medication management system for improving the medication adherence for patients, in order to save long term medication costs.

DETAILED DESCRIPTION:
Design, Setting and Patients: The investigators developed a mobile personalized medication management platform (PMMP) to reduce delayed and missed medications. The investigators conducted a randomized control trial in medical centers of northern Taiwan from January 2010 to July 2012 using 1198 participants that missed or delayed their medications during past three days. They received a minimum 7-day to 14-day maximum medication prescription.

Interventions: Patients were randomized into a control group which non-received any SMS reminder for medication using and an intervention group which received a SMS reminder everyday in mobile devices.

Primary Outcome(s) and Measure(s): The primary outcomes were compared patient medication adherence among experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Delayed or forgot to take medications over the last 3 days
* Received a min. 7-day medication prescription
* Able to receive SMS using mobile phones / devices
* 20 years or older
* Having intention to receive active treatment

Exclusion Criteria:

* Unable to receive SMS via mobile phones
* Illiterate and < 20 years of age
* Received outpatient prescription drugs for ≤ 7 days
* External use, injections and traditional Chinese medicine
* Planned to go abroad
* Cold, cough, or prescribed with analgesics

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in delaying and forgetting medications | Patients who participated in this trial will be sent SMS during 7days

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chuan Li, MD., PhD, Principal Investigator — Taipei Medical University

REFERENCES:
- [Derived] Huang CY, Nguyen PA, Clinciu DL, Hsu CK, Lu JR, Yang HC, Wu CC, Tsai WC, Chou YC, Kuo TBJ, Chang PL, Jian WS, Li YJ. A personalized medication management platform (PMMP) to improve medication adherence: A randomized control trial. Comput Methods Programs Biomed. 2017 Mar;140:275-281. doi: 10.1016/j.cmpb.2016.12.012. Epub 2016 Dec 30. PMID 28254084